CLINICAL TRIAL: NCT03650179
Title: Influence of the Urine Stream Interruption Exercise on the Micturition
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Gérard Amarenco, Head of Neuro-urology department, Tenon hospital, Pierre and Marie Curie University
Other Study IDs: P GREEN GRC 01
Record Dates: First submitted 2018-08-27; First posted 2018-08-28 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Voiding Function
Keywords: urine stream interruption exercise; voiding function; pelvic floor muscles exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients enrolled in the cohort: Patients over 18 years old, consulting for functional digestive disease, without neurologic or urologic disease, and performing an urodynamic examination in neuro-urology and functional explorations department.
  Interventions: Other: Observational study : No intervention

INTERVENTIONS:
Other: Observational study : No intervention — Observational study : No intervention. Only exporting data

SUMMARY:
This study assess micturition characteristic during and after a urine stream interruption exercise in patient without neurological or urologic disease.

DETAILED DESCRIPTION:
Urine stream interruption during voluntary voiding is often performed by women as a pelvic floor muscle exercise to develop urinary strength and avoid urinary incontinence. To our knowledge, there is no recommendation for performing urine stream interruption. Without evidence based data, stooping the urinary flow is reported as a risk of post void residual and urinary infection. The experts did not recommended to practice urine stream interruption as a pelvic floor exercise in urinary incontinence. However, during pelvic floor muscle training for urinary incontinence, exercises of urine stream interruption are often performed without knowledge of their consequences. The aim of this study is to assess micturition characteristic during and after a urine stream interruption exercise.

In this study, the investigators will compare the two uroflowmetries usually done in a Neuro-urology department of a University Hospital. Patient without neurological or urologic disease, consulting for a global evaluation of functional digestive disease and performing an urodynamic study will be included. During the urodynamic evaluation, two uroflowmetries are performed : one conventional uroflowmetry complying with the International Continence Society (ICS) recommendations and one uroflowmetry during exercise of urine stream interruption, as usually done in the department. Each uroflowmetry will be performed when the patient will feel a ''normal'' desire to void. For the urine stream interruption micturition, patients will be asked to "begin the micturition, stop at 3 seconds of micturition, when the stream is interrupt, start again voiding, again stop at 3 seconds of micturition and repeat this maneuver until the end of the micturition". As usual, sonographic estimation of post-void residual volume will complete each uroflowmetry.

The investigators will compare the voiding volume, the post-void residual volume, the maximal flow rate, the time to reach the maximal flow rate, the voiding time and the slope of the uroflowmetry (corresponding to the flow velocity acceleration) between the two uroflowmetries. For each voiding sequence of the urine stream interruption micturition the following parameters will be reported and compared: voiding volume and duration, maximal flow rate, time to reach the maximal flow rate, the latency to restart the micturition between each voiding sequence and the slope of the uroflowmetry.

Statistical analysis will be carried out using R 3.2.3 software (R Development Core Team, http://www.R-project.org) and R studio version 1.0.136. Differences between the two uroflowmetries will be evaluated using Student test. Correlation between the place of the voiding sequence in the urine stream interruption micturition and the different parameters will be evaluated using Pearson's correlations.

ELIGIBILITY:
Inclusion Criteria:

* follow in neuro-urology for functional digestive disease
* Appointment for urodynamic assessment

Exclusion Criteria:

* urological or neurological disease

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients consulting for an urodynamic assessment in a neuro-urology and functional explorations department
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
post-void residual volume | 1 Day : during the urodynamic assessment
  comparison between post-void residual volume during normal micturition and exercise of urine stream interruption

SECONDARY OUTCOMES:
maximal flow rate | 1 Day : during the urodynamic assessment
  comparison between maximal flow rate during normal micturition and exercise of urine stream interruption
time to reach the maximal flow rate | 1 Day : during the urodynamic assessment
  comparison between time to reach maximal flow rate during normal micturition and exercise of urine stream interruption
voiding time | 1 Day : during the urodynamic assessment
  comparison between the voiding time during normal micturition and exercise of urine stream interruption
the slope of the uroflowmetry (corresponding to the flow velocity acceleration) | 1 Day : during the urodynamic assessment
  comparison between the slope of the uroflowmetry during normal micturition and exercise of urine stream interruption

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PhD, Principal Investigator — GREEN GRC-01, Neuro-urology department, Hôpital Tenon
Locations (1):
- Department of Neuro-urology, Tenon hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No